CLINICAL TRIAL: NCT00120302
Title: Quality of Life Study in Adults With Facial Eczema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASM981CGB02
Record Dates: First submitted 2005-07-08; First posted 2005-07-15 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2008-01

CONDITIONS: Atopic Dermatitis
Keywords: Randomised; Placebo-controlled; Elidel; Quality of Life; Atopic Eczema
MeSH Terms: conditions — Dermatitis, Atopic | interventions — pimecrolimus

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Pimecrolimus
  Interventions: Drug: Pimecrolimus
- 2 (Placebo Comparator): Vehicle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pimecrolimus — Pimecrolimus cream 1 %
  Other Names: Elidel
  Arms: 1
Drug: Placebo — Matching vehicle cream
  Arms: 2

SUMMARY:
This study is not being conducted in the US.

The study consists of a 4 week double blind treatment period. All patients meeting the inclusion/exclusion criteria will enter the study at day 0 and be randomized into either pimecrolimus cream 1% or vehicle treatment groups in a 1:1 ratio. Patients will return to clinic on days 7,14 and 28 for assessments of disease severity. Patients who experience an unsatisfactory therapeutic effect, will attend an unscheduled visit and be withdrawn from the study.

Assessments of eligibility include an Investigator's Global Assessment and Pruritus score. Treatment history will be collected at baseline and Quality of Life Questionnaires will be carried out at every visit.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 years or older
* Active Moderate Facial AE at baseline (Facial IGA score of 3), within 3 days of a deterioration in symptoms that necessitates further treatment.
* Diagnosis of AE fulfilling the diagnostic criteria of Williams (Williams, et al. 1994) outlined below: *Must have an itchy skin condition plus 3 or more of the following 5 items listed below:

  1. History of involvement of the skin creases such as folds or elbows, behind the knees, fronts of ankles or around the neck;
  2. A personal history of asthma or hay fever;
  3. A history of a general dry skin in the last year;
  4. Visible flexural edema;
  5. Onset under the age of 2
* Pruritus score of 2 or above at baseline
* Patients in whom further use of TCS is clinically inappropriate due to:

  * burning, stinging, allergic reaction or other adverse event that prevents the patient from using topical corticosteroids to successfully treat an AE flare on the face;
  * presence of rosacea, telangiectasia, skin atrophy or glaucoma as a result of topical corticosteroid usage on the face;
  * presence of AE on the eyelids Or patients where previous treatment has been unsatisfactory and who would prefer to try an alternative treatment option.
* Patients who have been informed of the study procedures and have signed the informed consent form approved for the study. (Informed consent should be signed as instructed in ICH-GCP and local regulations).

Exclusion Criteria:

At baseline and throughout the study, females of childbearing potential:

* Who are pregnant or breast-feeding
* Who are menstruating, capable of becoming pregnant, and not practicing a medically approved method of contraception during and up to at least 4 weeks after the end of study treatment. A negative pregnancy test (urine) for all females of childbearing potential is required at the screening visit. 'Medically approved' contraception may include abstinence at the discretion of the investigator

At baseline and throughout the study, all patients:

* Who have received phototherapy (e.g. UVB, UVA) or systemic therapy (e.g. immunosuppressants, cytostatics) known or suspected to have an effect on AE within 1 month of Visit 1 (baseline)
* Who have received systemic corticosteroids (e.g. oral, intravenous, intra-articular, rectal) within 1 month of Visit 1. Patients on a stable maintenance dose of inhaled corticosteroids may participate
* Who have a known or suspected contact allergic dermatitis
* Who have received systemic antibiotics within 2 weeks prior to Visit 1.
* Who have used oral or topical antihistamines for the treatment of Pruritus within 2 weeks prior to visit 1
* Who have applied topical therapy (e.g. tar, topical corticosteroids, pimecrolimus or tacrolimus within 2 weeks prior to Screening
* Who have used potent or very potent TCS within 4 weeks prior to Visit 1.
* Who are immunocompromised (e.g. lymphoma, HIV infection/AIDS, Wiskott-Aldrich Syndrome) or have a history of malignant disease
* Who have a history of poor or no clinical response, or hypersensitivity to topical pimecrolimus cream 1%.
* Who have concurrent skin disease (e.g. acne) of such severity in the study area that it could interfere with the evaluation.
* Who have active bacterial (e.g. impetigo), viral (e.g. chicken pox, herpes simplex) or fungal infections (e.g. tinea corporis, intertriginosa)
* Who have received any investigational drugs within 8 weeks of visit 1, or plan to use any other investigational drugs during the course of this study
* Who, in the opinion of the investigator, are known to be unreliable, who are non-compliant with medical treatment, or are known to miss appointments
* Who have abuse problems, mental dysfunction or other factors limiting their ability to cooperate fully in study-related procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2005-03; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Change in quality of life score between baseline (study start) and week 4.

SECONDARY OUTCOMES:
Changes in patient's quality of life from baseline (study start) to 1 and 2 weeks after the beginning of treatment.
Between-treatment comparison of Investigator's Global Assessment (IGA) (face only); Patient's Global Assessment (face only); Pruritus (itch) Severity Assessment (face only).
Time from baseline (study start) to clearance of eczema.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (1):
- This study is not being conducted in the United States, Novartis Pharmaceuticals UK, Frimley, United Kingdom